CLINICAL TRIAL: NCT06545474
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) as an Early Intervention in Major Depression (MD) Compared to Antidepressant Selective Serotonin Reuptake Inhibitor (SSRI) Medication (Early-TMS)
Brief Title: Effects of rTMS Compared to SSRI as Early Treatment of Depression (Early-TMS)
Acronym: Early-TMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Center for Mental Health (DZPG; www.dzpg.org) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 614/2023BO1
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; non-invasive brain stimulation; repetitive transcranial magnetic stimulation; theta burst stimulation; non-treatment resistant depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- theta burst stimulation (TBS) (Experimental): In Stage I, participants receive 4-week bilateral theta burst stimulation. Bilateral TBS consists of 20 sessions that are conducted daily from Monday to Friday over a period of 4 weeks. The target regions are the right and left dorsolateral prefrontal cortex (dlPFC). On the left hemisphere, intermittent TBS (iTBS) is applied, which has a stimulating effect on the target region similar to 10 Hz rTMS. On the right dlPFC, continuous TBS (cTBS) is applied, which has an inhibitory effect similar to 1 Hz rTMS.
  Interventions: Device: bilateral theta burst stimulation
- SSRI treatment (Active Comparator): In Stage I, participants receive escitalopram (10mg/day) as standard medication for 4 weeks. In justified individual cases and according to the decision of the study physician, a higher dose or another SSRI can be administered.
  Interventions: Drug: SSRI treatment

INTERVENTIONS:
Device: bilateral theta burst stimulation — Each stimulation session consists of 600 stimuli applied in bursts of 3 pulses at 50 Hz, with an interstimulus interval of 200 ms. iTBS is administered 20 times for 2 seconds to the left dlPFC, with an intertrain interval of 8 seconds and cTBS continuously for 40 seconds to the right dlPFC in alternating order.
  Arms: theta burst stimulation (TBS)
Drug: SSRI treatment — Participants receive 4 weeks SSRI treatment with escitalopram (10mg/day) as standard drug.
  Arms: SSRI treatment

SUMMARY:
The aim of this randomized multicentre phase 2 clinical trial is to compare the effects of rTMS and SSRI medication as early treatment of depression. In this two-stage, therapy response-adapted trial, 106 patients suffering from non-treatment resistant major depression (non-TR MD) will be randomized in Stage I to either 4 weeks bilateral theta burst stimulation (TBS) or 4 weeks antidepressant SSRI medication. The allocation to Stage II occurs therapy response-adapted. Patients receive either a maintenance treatment or a switch to the respective other treatment arm. The primary outcome is the comparison of the two study arms with regard to therapy response measured with the Montgomery-Asberg Depression Rating Scale (MADRS) after 4 weeks at the end of Stage I.

DETAILED DESCRIPTION:
This is a therapy response-adapted, two-phase, randomized and controlled study. Initially, the study participants will be randomized to two treatment arms (Stage I: 4 weeks TBS vs. SSRI). After completion of Stage I, the allocation to Stage II (4 weeks) occurs therapy response-adapted. The type of further treatment depends on whether a remission, a treatment response or non-response has occurred in Stage I. If remission has been achieved, the treatment form already applied is continued as maintenance therapy. In the case of non-response, a switch to the other treatment arm takes place. For patients who show a treatment response but have not achieved remission, the corresponding patient preference is given special consideration for Stage II and thus determines the type of further treatment. Depending on patient preference, it is therefore possible both to continue treatment from Stage I and to switch to the other treatment arm.

The study aims to answer the question of whether a 4-week bilateral TBS is not inferior to standard antidepressant treatment with an SSRI in drug-naïve patients with MD in terms of efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* male, female, or diverse gender;
* age between 18 and 65 years;
* moderate to severe MD according to the diagnostic criteria of DSM-5;
* MADRS Score ≥ 20 points;
* the duration of the episode must be at least 2 weeks and not exceed a period of 2 years;
* no previous antidepressant treatment; indication for antidepressant medication;
* patients must be capable of giving informed consent.

Exclusion Criteria:

* acute suicidal ideation (MADRS item 10 score > 4);
* presence of psychotic symptoms;
* antiepileptic drugs or benzodiazepines in a dosage equivalent to > 1 mg Lorazepam/d;
* comorbid Axis I disorder (except anxiety disorders);
* presence of severe, clinically relevant, and predominant comorbid personality disorder;
* treatment resistance defined as the failure of at least one adequate antidepressant treatment attempt in the current or previous depressive episode;
* neurological pre-existing conditions such as severe traumatic brain injury, neoplasms, brain surgery, stroke within the last 3 months, neurodegenerative diseases: epilepsy or history of epileptic seizures;
* cardiac pacemaker (not compatible with MRI);
* intracranial metallic implants;
* previous rTMS treatment;
* deep brain stimulation;
* other severe somatic diseases; pregnancy;
* contraindications for the use of escitalopram.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
response rates after Stage I | 4 weeks
  The primary endpoint is the comparison of the two study arms with regard to the number of participants achieving therapy response (reduction of MADRS score ≥ 50%) after 4 weeks at the end of Stage I.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker-Sadzio J, Brendel B, Weller S, Bornheimer E, Mehlig U, Padberg F, Vogelmann U, Kammer T, Strube W, Martus P, Fallgatter AJ, Plewnia C. Effectiveness of rTMS compared to SSRI as early treatment of depression - study protocol of a randomized controlled trial (Early-TMS). Eur Arch Psychiatry Clin Neurosci. 2025 Sep;275(6):1839-1849. doi: 10.1007/s00406-025-01975-4. Epub 2025 Feb 22. PMID 39985658